CLINICAL TRIAL: NCT05082194
Title: The Relationship Between the Static and Dynamic Balance of the Body the Influence of Eyesight and Muscle Tension in the Cervical Spine in Cerebral Amyloid Angiopathy Patients - a Pilot Study
Brief Title: Balance Eyesight and Muscle Tension in the Cervical Spine in Cerebral Amyloid Angiopathy
Status: Completed | Type: Observational
Sponsor: Anna Olczak (Other)
Responsible Party: Sponsor-Investigator, Anna Olczak, PhD; Senior Specjalit of the Rehabilitation Clinc, Military Institute od Medicine National Research Institute
Organization: Military Institute od Medicine National Research Institute (Other)
Other Study IDs: 8/KRN/2020
Record Dates: First submitted 2021-09-30; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Cerebral Amyloid Angiopathy
Keywords: stroke,; CAA,; upper limb,; trunk exercises,; stabilization
MeSH Terms: conditions — Cerebral Amyloid Angiopathy; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Balance in CAA: Each of the examined post-stroke patients (CAA) performed the given test twice, with the eyes open the first time and the eyes closed the second time. Moreover, both during the Unterberger functional test and the tests on the Biodex SD balance platform, the muscle tone was assessed in the subjects using the Luna EMG device. In both tests, the patients performed each of the tests 6 times, 3 with eyes open and 3 with eyes closed, on the same day.
  Interventions: Procedure: balance with open and closed eyes
- Balance in healthy participants: Each of the examined healthy participants performed the given test twice, with the eyes open the first time and the eyes closed the second time. Moreover, both during the Unterberger functional test and the tests on the Biodex SD balance platform, the muscle tone was assessed in the subjects using the Luna EMG device. In both tests, the subject performed each of the tests 6 times, 3 with eyes open and 3 with eyes closed, on the same day.
  Interventions: Procedure: balance with open and closed eyes

INTERVENTIONS:
Procedure: balance with open and closed eyes — The UNTERBERGER TEST. The subjects performed the test once with their eyes open and then with their eyes closed. The participant's task was to assume a standing position with legs apart at hip-width and then walk in place (50 steps).
  Static and dynamic balance testing on the Biodex SD balance platform. Moreover, both during the Unterberger functional test and the tests on the Biodex SD balance platform, the muscle tone was assessed in the subjects using the Luna EMG device. Before starting the tests, surface electrodes were glued to the patient's body (according to the SENIAM procedure). Five surface electrodes were used, consisting of three channels. They were placed on the abdomen of the right sternocleidomastoid muscle, two more were placed on the left longus colli muscle, and one reference electrode on the right shoulder process of the scapula. After each completed test, an ongoing test report was generated.

SUMMARY:
Cerebral Amyloid Angiopathy (CAA) is one form of disease of the small vessels of the brain and can cause frequent cerebral hemorrhages as well as other types of stroke. The aim of the research was to examine the balance of the body in patients after a stroke and to determine how the tension of selected muscles of the cervical spine changes under the conditions of statics and dynamics, depending on the visual control or its absence.

DETAILED DESCRIPTION:
This is an observational study. The tests were performed with the use of tools and devices such as the Unterberger test, Biodex SD balance platform, and Luna EMG. The static equilibrium was assessed on a balance platform (stability test). The dynamic equilibrium was tested in the Unterberger test and on the balance platform (the fall risk test). All examinations were performed twice with eyes open and then closed. Additionally, during the tests, the tension of selected muscles of the cervical spine was recorded (the sternocleidomastoid muscle and the long neck muscle) (independent variables). It was examined how the intervention, static position, and dynamic displacement of the center of body mass, as well as the control and lack of eye control, influence the tension of selected muscles, and how the eyesight influences the body's balance in statics and dynamics (dependent variables). A group of healthy people was examined to assess whether neurological deficits in people after stroke could affect the results of static and dynamic balance and changes in muscle tone and whether the organ of vision plays a large role in controlling the center of body mass.

ELIGIBILITY:
Patients Inclusion Criteria:1) stroke in the course of CAA; 2) the functional state of the patients, which allows independent walking in a place and at a distance; 3) no severe deficits in communication, memory, or understanding what can impede proper measurement performance;

Patients Exclusion Criteria: 1) cause of stroke other than CAA; 2) stroke up to seven weeks after the episode; 3) epilepsy; 4) lack of trunk stability; 5) lack of independent walking; 6) high or very low blood pressure, dizziness, malaise.

Healthy Inclusion Criteria: 1) the control group consisted of healthy subjects with a stable trunk; 2) with independent walking.

Healthy Exclusion Criteria: 1) a history of neurologic or musculoskeletal disorders such as stroke or brain injury or other conditions that could affect their ability to active movement the trunk and the legs; 2) pain, dizziness; 3) permanent use of orthopedic supplies; 4) severe deficits in communication, memory, or understanding what can impede proper measurement performance; 5) high or very low blood pressure, dizziness, malaise.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study involved 8 patients after stroke in the course of Cerebral Amyloid Angiopathy (CAA) and 8 healthy subjects.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
static balance | up to 1 week
  TESTING STABILITY OF ATTITUDE with the use of the Biodex SD balance platform.
dynamic balance | up to 1 week
  FALL RISK TEST was assessed on the Biodex SD platform.
Unterberga Test | up to 1 week
  The subjects performed 50 steps, once with their eyes open and then with their eyes closed.
Sternocleidomastoid muscle tension | up to 1 week
  It was assessed on the Luna EMG
Longus Colli muscle tension | up to 1 week
  It was assessed on the Luna EMG

CONTACTS AND LOCATIONS:
Overall Officials: Anna Olczak, PhD, Principal Investigator — Military Institute of Medicine, Rehabilitation Clinic Poland
Locations (1):
- Military Institute of Medicine, Warsaw, Masovian District, Poland